CLINICAL TRIAL: NCT02651311
Title: Randomized Controlled Trial of the Postoperative Analgesic Efficacy of Ultrasound Guided Intermediate Cervical Plexus Block for Unipolar Sternocleidomastoid Release in Patient With Congenital Muscular Torticollis
Brief Title: Ultrasound Guided Intermediate Cervical Plexus Block for Congenital Muscular Torticollis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MED-DRU-15-002
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Muscular Torticollis
MeSH Terms: conditions — Congenital torticollis | interventions — Fentanyl; Ibuprofen

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block (Experimental): ultrasound guided intermediate cervical plexus block with 0.25% ropivacaine 0.2 ml/kg.
  Fentanyl in postanesthesia care unit(PACU), Ibuprofen in ward when pain scale (FLACC) is equal to or more than 4.
  Interventions: Other: intermediate cervical plexus block; Drug: Fentanyl; Drug: Ibuprofen
- No block (Placebo Comparator): Fentanyl in PACU, Ibuprofen in ward when pain scale (FLACC) is equal to or more than 4.
  Interventions: Drug: Fentanyl; Drug: Ibuprofen

INTERVENTIONS:
Other: intermediate cervical plexus block — ultrasound guided intermediate cervical plexus block with 0.25% ropivacaine 0.2 ml/kg
  Other Names: ultrasound guided intermediate cervical plexus block
  Arms: Block
Drug: Fentanyl — fentanyl 0.5 µg/kg in postanesthetic care unit when more or equal to FLACC scale 4.
Drug: Ibuprofen — ibuprofen in ward when more or equal to FLACC scale 4.

SUMMARY:
Congenital Muscular Torticollis (CMT) is a postural deformity of head and neck detected at birth or shortly after birth, primarily resulting from unilateral shortening of Sternocleidomastoid Muscle (SCM). Surgery could be chosen for the treatment for some children, which is accompanied by moderate pain and discomfort. The investigators focused the effectiveness of intermediates cervical plexus block because the dermatome of sensory of cervical plexus block is correlated to that of torticollis. So the effect of analgesia could decrease the use of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Undergoing general anesthesia for unipolar sternocleidomastoid release in patient with congenital muscular torticollis

Exclusion Criteria:

* coagulation disorder
* kidney or liver disease
* allergy to local anesthetics

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Pain on the FLACC scale | at 5 min after postanesthesia care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: yun jeong chae, Ph.D, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim JS, Joe HB, Park MC, Ahn H, Lee SY, Chae YJ. Postoperative Analgesic Effect of Ultrasound-Guided Intermediate Cervical Plexus Block on Unipolar Sternocleidomastoid Release With Myectomy in Pediatric Patients With Congenital Muscular Torticollis: A Prospective, Randomized Controlled Trial. Reg Anesth Pain Med. 2018 Aug;43(6):634-640. doi: 10.1097/AAP.0000000000000797. PMID 29781932